CLINICAL TRIAL: NCT07085572
Title: Cemiplimab as Maintenance Treatment for Advanced Adrenocortical Cancer
Acronym: INTERVAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Alfredo Berruti, Prof., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 6502; 2024-520449-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-16; First posted 2025-07-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-07

CONDITIONS: Adrenal Cortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cemiplimab added to the standard maintenance therapy with mitotane (Experimental)
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — 350 mg IV Q3W

SUMMARY:
This clinical trial is a single-arm, non-randomized, prospective phase II study.

The study aims to evaluate if the maintenance immunotherapy with cemiplimab in patients with AdrenoCortical Carcinoma (ACC), who obtained disease response or stabilization after first-line chemotherapy, may delay/prevent disease progression.

The study will be conducted at ASST Spedali Civili Hospital, Brescia - Italy.

DETAILED DESCRIPTION:
Adrenocortical carcinoma (ACC) is a rare malignancy affecting around 0.7-2 persons per one million population per year.

The only pharmacological approach approved by FDA and EMA for the treatment of ACC is mitotane, which has an adrenolytic effect causing adrenocortical insufficiency. So, the drug should be administered in association with glucocorticoid replacement for the purpose only of restoring the daily cortisol requirement.

Few therapeutic alternatives are available for metastatic ACC patients failing one to two lines of systemic treatment, so immunotherapy could represent a potential new treatment. The immune checkpoint inhibitors are the most promising immunotherapy agents in cancer pharmacology and have been also investigated in ACC. Bases on results of some clinical studies, immunotherapy has achieved long-term control in a small proportion of patients with metastatic ACC. We need to identify the patient subset destined to benefit most from this therapy and at what point in the therapeutic sequence of adrenal carcinoma should immunotherapy be introduced. We also need to implement strategies to overcome the intrinsic immuno-resistance of ACC.

The current strategy in the management of advanced ACC is the administration of the EDP (etoposide, doxorubicin, cisplatin) scheme associated with mitotane followed by maintenance mitotane in patients not progressing on chemotherapy. Maintenance immunotherapy could be administered in combination with mitotane, enhancing its efficacy. In addition, the powerful adrenolytic effect of mitotane could keep cortisol production inhibited, facilitating the efficacy of immunotherapy.

Maintenance therapy with cemiplimab in ACC patients after first-line chemotherapy may result in enhanced antitumor activity while avoiding potential interactions, including cross-resistance and cumulative toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females >18 years of age;
2. Patients with histologically confirmed ACC;
3. Previous induction therapy with EDP-M followed by cytoreductive surgery if indicated;
4. No disease progression after first line 4-6 EDP-M cycles;
5. An ECOG PS of 0, 1;
6. Adequate organ and bone marrow function documented by:

   1. Hemoglobin >9.0 g/dL
   2. ANC >1.5 x 109/L
   3. Platelet count >75 x 109/L
   4. Serum creatinine <1.5 ULN or estimated CrCl >30 mL/min
   5. Adequate hepatic function:

      * Total bilirubin <1.5 x ULN;
      * AST and ALT both <3 x ULN;
      * ALP <2.5 x ULN; Note: For patients with Gilbert's syndrome, total bilirubin ≤3x ULN. Gilbert's syndrome must be documented appropriately as past medical history.
7. Women of child-bearing potential (physiologically capable of becoming pregnant) that must agree to follow instructions for methods of contraception (including at least one highly effective contraception method, see study protocol) for the duration of treatment with study drug, and after discontinuation of treatment as long as mitotane plasma levels are detectable and, in any case, at least for 6 months post treatment completion; must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug;
8. Women must not be breastfeeding;
9. Males that must agree to follow instructions for methods of contraception (see study protocol) for the duration of treatment with study drug, and then for a total of 6 months post treatment completion. In addition, male patients must not donate sperm for the time period specified above;
10. Willing and able to comply with clinic visits and study-related procedures;
11. Willing and able to provide informed consent signed by study patient or legally acceptable representative;
12. Able to understand and complete study-related questionnaires.

Exclusion Criteria:

1. History of recent or active prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, breast ductal carcinoma in situ, or other treated malignancies where there has been no evidence of disease for at least 5 years;
2. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor;
3. Administration of a live vaccine within 30 days of the first dose of study treatment;
4. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs);
5. Diagnosis of immunodeficiency or systemic steroid therapy (i.e., dosing exceeding 10 mg of prednisone or equivalent). In case of mitotane treatment, a maximum steroid supplementation of 75 mg of cortone acetate (or equivalent hydrocortisone dose) will be accepted;
6. Uncontrolled HIV, Hepatitis B or Hepatitis C (see protocol for details);
7. History of (non-infectious) pneumonitis that required steroids or current pneumonitis;
8. Active infection requiring systemic therapy;
9. Significant cardiovascular disease, such as: history of myocardial infarction, acute coronary syndrome or coronary angioplasty / stenting / bypass grafting within the last 6 months OR CHF NYHA Class II-IV or history of CHF NYHA Class III or IV;
10. Pregnancy or breastfeeding;
11. Continued sexual activity in women of childbearing potential (physiologically capable of becoming pregnant) or sexually active men who are unwilling to practice highly effective contraception (including at least one highly effective contraception method, see study protocol) prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose;
12. History of active tuberculosis (TB, Bacillus Tuberculosis);
13. Untreated brain metastasis that may be considered active.
14. Known hypersensitivity or allergy to any of the excipients in the cemiplimab drug product.
15. Patients with a history of solid organ transplant (exception: corneal transplant)
16. Prior allogeneic stem cell transplantation, or autologous stem cell transplantation.
17. ECOG PS ≥ 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy of cemiplimab as a maintenance immunotherapy on PFS in patients with advanced ACC with no disease progression after 4-6 EDP-M cycles | 36 months
  Proportion of patients free from progression at 6 months after the end of first-line chemotherapy

SECONDARY OUTCOMES:
Evaluation of the effect of cemiplimab as a maintenance therapy on Overall Survival (OS) | 36 months
  The time from the date of the study start to the date of death due to any cause will be measured.
Evaluation of the effect of cemiplimab on patients' Quality of Life (QoL) | 36 months
  The QoL will be assesed by EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire) questionnaire.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Evaluation of the safety profile of maintenance cemiplimab therapy | 36 months
  The safety profile of maintenance cemiplimab therapy will be evaluated by the frequency of Adverse Effects (AEs) and laboratory abnormalities as graded by NCI CTCAE v5.0.

OTHER OUTCOMES:
Evaluation the safety of adding cemiplimab to standard mitotane therapy (Safety run-in phase) | At the end of Cycle 1 (each cycle is 21 days) for the first six patients enrolled.
  Frequency of occurrence of dose limiting toxicities (DLTs)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, Prof, MD, Principal Investigator — ASST Spedali Civili di Brescia and University of Brescia
Locations (1):
- S.C. Oncologia - ASST Spedali Civili di Brescia, Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powles T, Park SH, Caserta C, Valderrama BP, Gurney H, Ullen A, Loriot Y, Sridhar SS, Sternberg CN, Bellmunt J, Aragon-Ching JB, Wang J, Huang B, Laliberte RJ, di Pietro A, Grivas P. Avelumab First-Line Maintenance for Advanced Urothelial Carcinoma: Results From the JAVELIN Bladder 100 Trial After >/=2 Years of Follow-Up. J Clin Oncol. 2023 Jul 1;41(19):3486-3492. doi: 10.1200/JCO.22.01792. Epub 2023 Apr 18. PMID 37071838
- [Background] Powles T, Park SH, Voog E, Caserta C, Valderrama BP, Gurney H, Kalofonos H, Radulovic S, Demey W, Ullen A, Loriot Y, Sridhar SS, Tsuchiya N, Kopyltsov E, Sternberg CN, Bellmunt J, Aragon-Ching JB, Petrylak DP, Laliberte R, Wang J, Huang B, Davis C, Fowst C, Costa N, Blake-Haskins JA, di Pietro A, Grivas P. Avelumab Maintenance Therapy for Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2020 Sep 24;383(13):1218-1230. doi: 10.1056/NEJMoa2002788. Epub 2020 Sep 18. PMID 32945632
- [Background] Cosentini D, Grisanti S, Dalla Volta A, Lagana M, Fiorentini C, Perotti P, Sigala S, Berruti A. Immunotherapy failure in adrenocortical cancer: where next? Endocr Connect. 2018 Dec;7(12):E5-E8. doi: 10.1530/EC-18-0398. PMID 30400026
- [Background] Le Tourneau C, Hoimes C, Zarwan C, Wong DJ, Bauer S, Claus R, Wermke M, Hariharan S, von Heydebreck A, Kasturi V, Chand V, Gulley JL. Avelumab in patients with previously treated metastatic adrenocortical carcinoma: phase 1b results from the JAVELIN solid tumor trial. J Immunother Cancer. 2018 Oct 22;6(1):111. doi: 10.1186/s40425-018-0424-9. PMID 30348224
- [Background] Klein O, Senko C, Carlino MS, Markman B, Jackett L, Gao B, Lum C, Kee D, Behren A, Palmer J, Cebon J. Combination immunotherapy with ipilimumab and nivolumab in patients with advanced adrenocortical carcinoma: a subgroup analysis of CA209-538. Oncoimmunology. 2021 Apr 12;10(1):1908771. doi: 10.1080/2162402X.2021.1908771. PMID 33889439
- [Background] McGregor BA, Campbell MT, Xie W, Farah S, Bilen MA, Schmidt AL, Sonpavde GP, Kilbridge KL, Choudhury AD, Mortazavi A, Shah AY, Venkatesan AM, Bubley GJ, Siefker-Radtke AO, McKay RR, Choueiri TK. Results of a multicenter, phase 2 study of nivolumab and ipilimumab for patients with advanced rare genitourinary malignancies. Cancer. 2021 Mar 15;127(6):840-849. doi: 10.1002/cncr.33328. Epub 2020 Nov 20. PMID 33216356
- [Background] Carneiro BA, Konda B, Costa RB, Costa RLB, Sagar V, Gursel DB, Kirschner LS, Chae YK, Abdulkadir SA, Rademaker A, Mahalingam D, Shah MH, Giles FJ. Nivolumab in Metastatic Adrenocortical Carcinoma: Results of a Phase 2 Trial. J Clin Endocrinol Metab. 2019 Dec 1;104(12):6193-6200. doi: 10.1210/jc.2019-00600. PMID 31276163
- [Background] Bedrose S, Miller KC, Altameemi L, Ali MS, Nassar S, Garg N, Daher M, Eaton KD, Yorio JT, Daniel DB, Campbell M, Bible KC, Ryder M, Chintakuntlawar AV, Habra MA. Combined lenvatinib and pembrolizumab as salvage therapy in advanced adrenal cortical carcinoma. J Immunother Cancer. 2020 Jul;8(2):e001009. doi: 10.1136/jitc-2020-001009. PMID 32737143
- [Background] Habra MA, Stephen B, Campbell M, Hess K, Tapia C, Xu M, Rodon Ahnert J, Jimenez C, Lee JE, Perrier ND, Boraddus RR, Pant S, Subbiah V, Hong DS, Zarifa A, Fu S, Karp DD, Meric-Bernstam F, Naing A. Phase II clinical trial of pembrolizumab efficacy and safety in advanced adrenocortical carcinoma. J Immunother Cancer. 2019 Sep 18;7(1):253. doi: 10.1186/s40425-019-0722-x. PMID 31533818
- [Background] Naing A, Meric-Bernstam F, Stephen B, Karp DD, Hajjar J, Rodon Ahnert J, Piha-Paul SA, Colen RR, Jimenez C, Raghav KP, Ferrarotto R, Tu SM, Campbell M, Wang L, Sabir SH, Tapia C, Bernatchez C, Frumovitz M, Tannir N, Ravi V, Khan S, Painter JM, Abonofal A, Gong J, Alshawa A, McQuinn LM, Xu M, Ahmed S, Subbiah V, Hong DS, Pant S, Yap TA, Tsimberidou AM, Dumbrava EEI, Janku F, Fu S, Simon RM, Hess KR, Varadhachary GR, Habra MA. Phase 2 study of pembrolizumab in patients with advanced rare cancers. J Immunother Cancer. 2020 Mar;8(1):e000347. doi: 10.1136/jitc-2019-000347. PMID 32188704
- [Background] Grisanti S, Cosentini D, Lagana M, Volta AD, Palumbo C, Massimo Tiberio GA, Sigala S, Berruti A. The long and winding road to effective immunotherapy in patients with adrenocortical carcinoma. Future Oncol. 2020 Dec;16(36):3017-3020. doi: 10.2217/fon-2020-0686. Epub 2020 Aug 28. No abstract available. PMID 32857613
- [Background] Raj N, Zheng Y, Kelly V, Katz SS, Chou J, Do RKG, Capanu M, Zamarin D, Saltz LB, Ariyan CE, Untch BR, O'Reilly EM, Gopalan A, Berger MF, Olino K, Segal NH, Reidy-Lagunes DL. PD-1 Blockade in Advanced Adrenocortical Carcinoma. J Clin Oncol. 2020 Jan 1;38(1):71-80. doi: 10.1200/JCO.19.01586. Epub 2019 Oct 23. PMID 31644329
- [Background] Cremaschi V, Abate A, Cosentini D, Grisanti S, Rossini E, Lagana M, Tamburello M, Turla A, Sigala S, Berruti A. Advances in adrenocortical carcinoma pharmacotherapy: what is the current state of the art? Expert Opin Pharmacother. 2022 Aug;23(12):1413-1424. doi: 10.1080/14656566.2022.2106128. Epub 2022 Aug 3. PMID 35876101
- [Background] Fassnacht M, Assie G, Baudin E, Eisenhofer G, de la Fouchardiere C, Haak HR, de Krijger R, Porpiglia F, Terzolo M, Berruti A; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Adrenocortical carcinomas and malignant phaeochromocytomas: ESMO-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Nov;31(11):1476-1490. doi: 10.1016/j.annonc.2020.08.2099. Epub 2020 Aug 27. No abstract available. PMID 32861807
- [Background] Berruti A, Baudin E, Gelderblom H, Haak HR, Porpiglia F, Fassnacht M, Pentheroudakis G; ESMO Guidelines Working Group. Adrenal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii131-8. doi: 10.1093/annonc/mds231. No abstract available. PMID 22997446